CLINICAL TRIAL: NCT03467633
Title: Atrial Fibrillation Trial to Evade Recurrence: effectS of Hiit Before electrO-Cardioversion
Brief Title: Atrial Fibrillation Trial to Evade Recurrence: effectS of Hiit Before electrO-Cardioversion for 3-weeKs
Acronym: AFTERSHOCK
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough participants recruited.
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Cardiac Arrhythmia Network of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20170868
Record Dates: First submitted 2018-02-13; First posted 2018-03-16 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity interval training (HIIT) (Experimental): Participants in the HIIT group will receive 3-weeks of tri-weekly supervised exercise sessions at the University of Ottawa Heart Institute prior to their scheduled electro-cardioversion. The session will last 23 minutes in duration and consist of a 2-minute warm-up at 50% of peak power output (PPO), 2 x 8-minute interval training blocks of 30 seconds at 80-100% of PPO interspersed with 30-seconds of active recovery and a 1-minute cool down at 25 % of PPO. The sessions will be lead by a Registered Kinesiologist.
  Interventions: Behavioral: High-intensity interval training
- Usual Care Control (No Intervention): Participants assigned to the control group will have usual care, which involves no behavioural interventions leading up to their electro-cardioversion.

INTERVENTIONS:
Behavioral: High-intensity interval training — Participants in the HIIT group will receive 3-weeks of tri-weekly supervised exercise sessions at the UOHI prior to their scheduled electro-cardioversion. The session will last 23 minutes in duration and consist of a 2-minute warm-up at 50% of peak power output (PPO), 2 x 8-minute interval training blocks of 30 seconds at 80-100% of PPO interspersed with 30-seconds of active recovery and a 1-minute cool down at 25 % of PPO. The sessions will be lead by a Registered Kinesiologist.
  Arms: High-intensity interval training (HIIT)

SUMMARY:
This is a study looking at the feasibility of conducting a larger definitive research trial looking at the effectiveness of high intensity interval training in individuals who are scheduled for electro-cardioversion. Usual care for these participants is to go home and continue with their typical daily routine. The investigators will test whether participating in 3-weeks of thrice-weekly high intensity interval training before electro-cardioversion can lengthen the time to recurrence of atrial fibrillation after electro-cardioversion in these individuals. Participants will be asked to come to the University of Ottawa Heart Institute for a baseline visit at which fitness (cycle ergometer), body composition (weight, height, waist circumference and percentage body fat), heart rate variability and habitual exercise levels will be measured. Participants will then be randomized to either the exercise group or the usual care group. Those randomized to the usual care group will go home for 3-weeks and continue with their typical daily routine. Those randomized to the exercise group will return to the Heart Institute three times per week for 3-weeks to participate in a high intensity interval training program prior to their electro-cardioversion. All participants will be asked to measure daily heart rate and rhythm using the AliveCor system which is compatible with their Smartphones, for up to 12-months following their electro-cardioversion. All participants will be asked to return at 3-weeks (and prior to their electro-cardioversion) to measure fitness (cycle ergometer), body composition (weight, height, waist circumference and percentage body fat), and habitual exercise levels. The entire study should last approximately 24-months. Participants will be involved for 52-weeks. The investigators are looking to recruit 20 participants total for the feasibility trial. The investigators hypothesize that recruitment rates, drop-out rates, and adherence to the intervention will support a larger definitive trial.

DETAILED DESCRIPTION:
This is a study looking at the feasibility of conducting a larger definitive research trial looking at the effectiveness of high intensity interval training on lengthening time to recurrence of persistent atrial fibrillation in individuals who are scheduled for electro-cardioversion. Usual care for these participants is to go home and continue with their typical daily routine until their scheduled cardioversion. The investigators will test whether participating in 3-weeks of thrice-weekly high intensity interval training before electro-cardioversion can lengthen the time to recurrence of atrial fibrillation after electro-cardioversion in these individuals. Participants will be asked to come to the University of Ottawa Heart Institute for a baseline visit at which fitness (cycle ergometer), body composition (weight, height, waist circumference and percentage body fat), and habitual exercise levels will be measured. Participants will then be randomized to either the exercise group or the usual care group. Those randomized to the usual care group will go home for 3-weeks and continue with their typical daily routine. Those randomized to the exercise group will return to the Heart Institute three times per week for 3-weeks to participate in a high intensity interval training cycle ergometer program prior to their electro-cardioversion. All participants will be asked to return at 3-weeks (and prior to their electro-cardioversion) to measure fitness (cycle ergometer), body composition (weight, height, waist circumference and percentage body fat), and habitual exercise levels. Following the electro-cardioversion, all participants will be asked to measure daily heart rate and rhythm using the AliveCor system which is compatible with their Smartphones/tablets/iPads, for up to 12-months or until they return to persistent atrial fibrillation. The entire study should last approximately 24-months. Participants will be involved for a maximum of 52-weeks. The investigators are looking to recruit a total of 20 participants for the feasibility trial. The investigators hypothesize that recruitment rates, drop-out rates, and adherence to the intervention will support a larger definitive trial.

ELIGIBILITY:
Inclusion Criteria:

1. Persistent atrial fibrillation
2. Eligible and scheduled for electro-cardioversion at UOHI
3. Rate controlled with a resting ventricular rate of equal to or less than 100bpm
4. Between 18-85 years of age
5. Owns a Smartphone
6. Physically able to participate in exercise
7. Willing and able to provide written, informed consent
8. Willing and able to return for follow-up visits
9. Willing and able to provide daily ECG recordings using the AliveCor system for the duration of the study.

Exclusion Criteria:

1. Participating in routine exercise training (more than two times per week) in the past 3 months
2. Atrial Flutter secondary to ablation
3. Unstable angina
4. Diagnosed with severe mitral or aortic stenosis, hypertrophic obstructive cardiomyopathy
5. Pregnant, lactating or planning to become pregnant during the study period
6. Diagnosed with rheumatic heart disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2020-10-08 (Actual)

PRIMARY OUTCOMES:
Feasibility - recruitment rates | 52-weeks
  recruitment rates
Feasibility - loss to follow-up and drop-out rates | 52-weeks
  loss to follow-up and drop-out rates
Feasibility - reasons for drop-out | 52-weeks
  reasons for drop-out
Feasibility - adherence to study procedures | 52-weeks
  adherence to study procedures including daily AliveCor measures
Feasibility - attendance at thrice-weekly HIIT sessions | 3-weeks
  attendance at thrice-weekly HIIT sessions

SECONDARY OUTCOMES:
Time to recurrence of atrial fibrillation | Up to 52 weeks after electro-cardioversion.
  Time to recurrence will be measured with a daily ECG recording up to 52-weeks from randomization, using the AliveCor system and Smartphone.
Physical Activity levels | 3-weeks
  Participants will also be asked to complete a questionnaire related to habitual physical activity (modified Godin) at baseline and follow-up. The modified Godin asks participants to recall the last 7 days and report the number of days and the number of minutes per day they participated in mild, moderate and vigorous bouts of physical activity. These values are then multiplied together to calculate minutes/week of mild physical activity and minutes/ week of moderate-to-vigorous intensity physical activity.
Fitness | 3-weeks
  Participants will complete a CPET at baseline and 3-weeks to assess fitness level using a pre-determined protocol on a cycle ergometer (Oxycon mobile, CareFusion, USA).
Clinical outcomes | 3-weeks
  Body composition will be assessed: height
Weight | 3-weeks
  Body composition will be assessed: weight
Waist Circumference | 3-weeks
  Body composition will be assessed: waist circumference
Body Mass Index | 3-weeks
  Body composition will be assessed: body mass index
Body Fat | 3-weeks
  Body composition will be assessed:body fat percentage

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Reed, PhD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No